CLINICAL TRIAL: NCT06395012
Title: A Phase 1, Randomized, Placebo-controlled, Investigator and Participant Blinded, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of LY3985297 in Healthy Participants
Brief Title: A First-In-Human Study of LY3985297 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18794; J4S-MC-KSAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: LY3985297 (Cohorts 1-8) (Experimental): Single ascending dose of LY3985297 administered either intravenously (IV) or subcutaneously (SC). Cohort 5,6 and 7 is conducted in Japanese or Chinese participants.
  Interventions: Drug: LY3985297
- Part B: LY3985297 (Cohorts 1-4) (Experimental): Multiple ascending dose of LY3985297 administered either IV or SC.
  Interventions: Drug: LY3985297
- Placebo Comparator: Part A and B: Placebo (Placebo Comparator): Placebo administered either IV or SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3985297 — Administered either IV or SC.
  Arms: Part A: LY3985297 (Cohorts 1-8); Part B: LY3985297 (Cohorts 1-4)
Drug: Placebo — Administered either IV or SC.
  Arms: Placebo Comparator: Part A and B: Placebo

SUMMARY:
The main purpose of this study is to see if LY3985297, the study drug, is safe and well-tolerated when given as a single dose or as multiple doses either through an intravenous (into a vein) or a subcutaneous (under the skin) injection in healthy participants. Study will also evaluate how much of the study drug LY3985297 gets into the blood stream and how long it takes the body to remove it.

The study is conducted in two parts (part A and B), each part has a separate treatment cohort.

The study will last up to approximately 116 days for part A, and 145 days for part B, including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be overtly healthy, as determined by medical evaluation.
* Have a body mass index of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive, and a minimum body weight of 45.0 kg.
* Participants must be assigned male or female at birth and not of childbearing potential.
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), clinical laboratory test results that are acceptable for the study.
* Have venous access sufficient to allow for blood sampling.

For Part A Cohorts 5, 6, and 7:

* Participants must be first-generation Japanese only, defined as the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Japanese descent and born in Japan. Or
* Participants must be first-generation Chinese only, defined as the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Chinese descent and born in China.

Exclusion Criteria:

* Have a current or recent acute, active infection. For at least 30 days before screening and up to the randomization visit (Day 1).
* Had any surgical procedure (except for minor surgery requiring local or no anesthesia and without any complications or sequelae) within 12 weeks prior to screening or intend to during the study.
* Have a history of multiple or severe allergies, or an anaphylactic reaction, to prescription or nonprescription drugs or food.
* Show evidence of active or latent tuberculosis (TB).
* Have one of the following infections: hepatitis B, C virus or human immunodeficiency virus (HIV).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration | Baseline up to Week 13 (Part A), Week 17 (Part B)
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3985297 following intravenous (IV) administration | Predose on day 1 up to Week 13 (Part A), Week 17 (Part B)
PK: Cmax of LY3985297 following subcutaneous (SC) administration | Predose on day 1 up to Week 13 (Part A), Week 17 (Part B)
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3985297 following IV administration | Predose on day 1 up to Week 13 (Part A), Week 17 (Part B)
PK: AUC of LY3985297 following SC administration | Predose on day 1 up to Week 13 (Part A), Week 17 (Part B)
Bioavailability (%F) of LY3985297 following SC administration | Predose on day 1 up to Week 13 (Part A), Week 17 (Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - CenExel ACT, Anaheim, California
  - ICON, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No